CLINICAL TRIAL: NCT02752672
Title: Study on the Therapeutic Mechanisms of Dithranol Treatment With Regard to Pro- and Contra-inflammatory Factors, microRNA as Well as Lymph and Blood Vessels in Patients With Chronic Plaque Psoriasis
Brief Title: Study on the Therapeutic Mechanisms of Dithranol Treatment in Patients With Chronic Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Klinikum Klagenfurt am Wörthersee (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Univ.Prof. Dr. Peter Wolf, Medical University of Graz
Other Study IDs: A 23/15
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Psoriasis
Keywords: dithranol; therapeutic mechanisms
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis: Psoriasis patients treated with dithranol
- Non-Psoriasis: Non-Psoriasis patients undergoing surgery for skin lesions. Tumor-adjacent skin is collected for control purposes.

SUMMARY:
Dithranol (known in the U.S.A. as anthralin and in Germany as cignolin) is one of the oldest and safest topical anti-psoriatic treatments. However, despite explorative investigations, the skin disease-clearing mechanisms of dithranol remain poorly understood (Painsi et al, JDDG 2015). The purpose of this study is to investigate the therapeutic mechanisms of dithranol in psoriasis.

DETAILED DESCRIPTION:
Skins biopsies from psoriatic skin and blood samples will be taken before (day 0) and at several time points after start (day 4, week 2-3, and week 6-7) of dithranol therapy to be subjected to an explorative analysis (see outcome measures). A total of maximal 15 psoriasis patients will be enrolled. Normal lesion-adjacent skin from 10 patients undergoing surgery for non-inflammatory conditions will serve as control.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years of age
* Clinical diagnosis of chronic plaque psoriasis
* Dithranol treatment scheduled

Exclusion Criteria:

* Systemic anti-psoriatic therapy (DMARD, phototherapy and/or Biologics) within 4 weeks of study entry (start of dithranol treatment)
* Topical treatment with steroids and or vitamin D3 analogues within 2 weeks of study entry (start of dithranol treatment)
* Autoimmune disorders
* Poor general health status
* Intolerance of dithranol
* Pregnancy and lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of maximal 15 psoriasis patients will be enrolled. Normal lesion-adjacent skin from 10 patients undergoing surgery for non-inflammatory conditions will serve as control.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Protein and mRNA expression of pro- and contra-inflammatory factors in the skin and blood | day 0, 4, 14, 42

SECONDARY OUTCOMES:
MicroRNA expression in skin and blood | day 0, 4, 14, 42
Size and density of lymph and blood vessels in the skin | day 0, 4, 14, 42
Angiogenic factors and their receptors in the skin | day 0, 4, 14, 42
Inflammatory infiltrate in the skin and alterations of the epidermis | day 0, 4, 14, 42
Microarray analysis of skin samples and subsequent targeted analysis of deregulated genes | day 0, 4, 14, 42

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Klagenfurt am Woerthersee, Klagenfurt, Carinthia, Austria

REFERENCES:
- [Derived] Graier T, Golob-Schwarzl N, Weger W, Benezeder T, Painsi C, Salmhofer W, Wolf P. Furin Expression in Patients With Psoriasis-A Patient Cohort Endangered to SARS-COV2? Front Med (Lausanne). 2021 Feb 10;8:624462. doi: 10.3389/fmed.2021.624462. eCollection 2021. PMID 33644099
- [Derived] Benezeder T, Painsi C, Patra V, Dey S, Holcmann M, Lange-Asschenfeldt B, Sibilia M, Wolf P. Dithranol targets keratinocytes, their crosstalk with neutrophils and inhibits the IL-36 inflammatory loop in psoriasis. Elife. 2020 Jun 2;9:e56991. doi: 10.7554/eLife.56991. PMID 32484435